CLINICAL TRIAL: NCT06552546
Title: Pharmacokinetics of Single- and Double-dose Icodextrin in Patients on Peritoneal Dialysis
Brief Title: Pharmacokinetics of Single- and Double-dose Icodextrin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Professor, Peking University First Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-524
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Peritoneal Dialysis
Keywords: Icodextrin; Pharmacokinetics; Peritoneal dialysis
MeSH Terms: interventions — Icodextrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SICO(single-dose icodextrin) (Experimental): Eligible participants used one icodextrin bag (single-dose icodextrin, SICO) on the first day. Icodextrin solution was left in the peritoneal cavity for a 8-hour dwell. After the icodextrin exchange, the solution was drained from the peritoneal cavity and the patients resumed dialysis using dextrose dialysate with three additional manual exchanges performed for the balance of the 24 hours since the icodextrin dwell was initiated. Patients were discharged and requested to return on days 7 and 14. Blood, urine and dialysate samples are collected at the time-points as required. Icodextrin and metabolites were analyzed and the pharmacokinetics profiles of single-dose icodextrin were provided.
  Interventions: Drug: Icodextrin
- DICO(double-dose icodextrin) (Experimental): Eligible participants used two icodextrin bags (double-dose icodextrin, DICO) on the first day. Each icodextrin solution was left in the peritoneal cavity for a 8-hour dwell. The double-dose icodextrin was administered in a sequential way. After the icodextrin exchange, the solution was drained from the peritoneal cavity and the patients resumed dialysis using dextrose dialysate with three additional manual exchanges performed for the balance of the 24 hours since the icodextrin dwell was initiated. Patients were discharged and requested to return on days 7 and 14. Blood, urine and dialysate samples are collected at the time-points as required. Icodextrin and metabolites were analyzed and the pharmacokinetics profiles of double-dose icodextrin were provided.
  Interventions: Drug: Icodextrin

INTERVENTIONS:
Drug: Icodextrin — Eligible participants were admitted to the hosptial ward and used one icodextrin bag (single-dose icodextrin) or two icodextrin bags (double-dose icodextrin) on the first day, depending on their choice. Each icodextrin solution was left in the peritoneal cavity for a 8-hour dwell. The double-dose icodextrin was administered in a sequential way. After the icodextrin exchange(s), the solution was drained from the peritoneal cavity and the patients resumed dialysis using dextrose dialysate with two or three additional manual exchanges performed for the balance of the 24 hours since the icodextrin dwell was initiated. Patients were discharged and requested to return on days 7 and 14. Blood, urine and dialysate samples are collected at the time-points as required. Icodextrin and metabolites were analyzed and the pharmacokinetics profiles of single- and double-dose icodextrin were provided.
  Other Names: Extraneal®，Baxter Healthcare (Guangzhou) Co., Ltd.， Guangzhou，China

SUMMARY:
The study aims to provide the pharmacokinetics profiles of single- and double-dose icodextrin in patients on peritoneal dialysis (PD). It may expand the available knowledge of the clinical pharmacology of icodextrin following its intraperitoneal administration and fills the gaps in our understanding of the fate of icodextrin and the metabolic consequences of icodextrin and its metabolites.

DETAILED DESCRIPTION:
Icodextrin is confirmed safe and effective as an alternative osmotic agent by numerous clinical studies. Due to its high molecular weight, icodextrin exerts its effect to enhance ultrafiltration (UF) during long (10~14 hours) dwells through prolonged colloid osmosis across the peritoneal membrane in PD patients. However, the utilization of icodextrin is currently limited to 1 exchange per day in order to avoid plasma accumulation of maltose or other metabolites. Two icodextrin bags per day has been reported to be safely prolong PD technique survival in patients in whom one icodextrin exchange provides insufficient UF. A detailed evaluation of the pharmacokinetics and elimination of icodextrin and metabolites following a single exchange has been reported. However, characterization of the plasma kinetics, metabolism and elimination of double dose icodextrin is not available yet. Therefore, we design the study to provide the pharmacokinetics profile of single- and double-dose icodextrin in patients on peritoneal dialysis. It may expand the available knowledge of the clinical pharmacology of icodextrin following its intraperitoneal administration and fills the gaps in our understanding of the fate of icodextrin and the metabolic consequences of icodextrin and its metabolites.

Eligible participants were admitted to the hosptial ward and used one icodextrin bag (single-dose icodextrin) or two icodextrin bags (double-dose icodextrin) on the first day, depending on their choice. Each icodextrin solution was left in the peritoneal cavity for a 8-hour dwell. The double-dose icodextrin was administered in a sequential way. After the icodextrin exchange(s), the solution was drained from the peritoneal cavity and the patients resumed dialysis using dextrose dialysate with two or three additional manual exchanges performed for the balance of the 24 hours since the icodextrin dwell was initiated. Patients were discharged and requested to return on days 7 and 14. Blood, urine and dialysate samples are collected at the time-points as required. Icodextrin and metabolites were analyzed and the pharmacokinetics profiles of single- and double-dose icodextrin were provided.

Icodextrin was quantified in plasma, urine and dialysate by exhaustive hydrolysis of all glucose polymers to glucose using the enzyme amyloglucosidase. Free glucose (determined prior to hydrolysis) was subtracted from the result of hydrolysis to obtain the icodextrin concentration. Maltose (DP2), maltotriose (DP3), maltotetraose (DP4) were individually quantified in blood, spent dialysate and urine (for patients with urine output) using liquid chromatography-tandem mass spectrometry (LC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease, receiving peritoneal dialysis for > 3 months, and clinically stable.
* Suitable for 4 exchanges of manual peritoneal dialysis on the first study day.

Exclusion Criteria:

* History of allergic reaction to icodextrin dialysis solution or corn starch;
* With malignant tumor receiving radiotherapy and/or chemotherapy, active hepatitis or hepatic failure, active autoimmune disease, severe digestive malabsorption or an eating disorder, or HIV/AIDS;
* Acute systemic infection, peritonitis, catheter-related infection, cardiovascular disease, surgery, or trauma in the previous one month;
* A high probability of receiving a kidney transplant or transferring to hemodialysis or drop-out due to socioeconomic causes within 1 months;
* Receiving hybrid dialysis (peritoneal dialysis combined with hemodialysis);
* Pregnant or lactating female;
* Having used icodextrin within previous 30 days；
* Peritoneal catheter dysfunction；
* Not suitable for enrollment assessed by researchers, including those unable followed the study protocol, or enrolled in other intervention studies, or with other reasons considering not suitable for enrollment by researchers.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | SICO: 0, 4, 8, 10, 12,16, 20, 24, 48, 72 hour, and day 7 and 14; DICO: 0, 4, 8, 12,16, 18, 20, 24, 28, 32, 56, 80 hour and day 7 and 14
  The maximum serum concentration of icodextrin that occurs after administration.
Peak time (Tmax) | SICO: 0, 4, 8, 10, 12,16, 20, 24, 48, 72 hour, and day 7 and 14; DICO: 0, 4, 8, 12,16, 18, 20, 24, 28, 32, 56, 80 hour and day 7 and 14
  Time (hours) to achieve the maximum serum concentration.
Area under the concentration-time curve（AUC） | 14 days
  AUC based on icodextrin serum concentrations.
Elimination half life（t1/2） | 14 days
  How long it takes for blood levels to drop by half. This parameter directly reflects the rate at which the drug is eliminated from the body.
Clearance(CL) | 14 days
  Serum icodextrin clearance.

SECONDARY OUTCOMES:
Adverse Events | 14 days
  Any adverse events throughout entirety of study as assessed by physician investigator

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Professor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No